CLINICAL TRIAL: NCT07049055
Title: A Phase I/IIa Randomized Clinical Trial to Evaluate the Efficacy of EGFR-targeted, PNU-159682-packaged Nanocells & Glycolipid-Packaged Nanocells in Combination With Gemcitabine & Nab-paclitaxel in Metastatic Pancreatic Ductal Adenocarcinoma
Brief Title: A Clinical Trial to Evaluate EDV Nanocell Therapy With Gemcitabine and Nab-paclitaxel in Pancreatic Cancer
Acronym: Carolyn-USA
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Engeneic Pty Limited (Industry)
Collaborators: Herbert Irving Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ENG15
Record Dates: First submitted 2025-05-29; First posted 2025-07-03 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Pancreatic Cancer, Metastatic; PDAC - Pancreatic Ductal Adenocarcinoma
Keywords: PDAC; Molecular Targeted Therapy; Drug Delivery Systems; Pancreatic Cancer; Epidermal Growth Factor Receptor; Bispecific Antibodies; Antineoplastic Agents; Immunotherapy; Disease Progression
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasm Metastasis; Disease Progression | interventions — Gemcitabine; Taxes

STUDY DESIGN:
Intervention Model Description: This is a randomized blinded Phase I/IIa study to test the safety and efficacy of E-EDV-D682/GC in combination with gemcitabine and nab-paclitaxel.
  The study design is based on an initial safety run-in using a rolling 6 model prior to randomization into two treatment arms. The initial safety run-in (Cohort I) will assess safety and tolerability of E-EDV-D682/GC in combination with gemcitabine and nab-paclitaxel in subjects with metastatic PDAC. In Cohort 2 subjects will be randomized into two treatment arms consisting of E-EDV-D682/GC with gemcitabine and nab-paclitaxel or gemcitabine and nab-paclitaxel with placebo.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 2 Arm A (Experimental): E-EDV-D682/GC with gemcitabine and nab-paclitaxel
  Interventions: Drug: E-EDV-D682; Drug: EDV-GC; Drug: Gemcitabine; Drug: Nab paclitaxel.
- Cohort 2 Arm B (Placebo Comparator): gemcitabine and nab-paclitaxel with placebo
  Interventions: Drug: Gemcitabine; Drug: Nab paclitaxel.

INTERVENTIONS:
Drug: E-EDV-D682 — E-EDV-D682 is a product based on the EnGeneIC EDV™ technology. EDVs are bacterially derived nanocells 400 nm in diameter that can be packaged with a range of different chemotherapeutic drugs and specifically targeted to cancer cell receptors via single chain bispecific antibodies (BsAb).
  E-EDV-D682 packages a chemotherapeutic payload PNU159682 into the EDV which targets the epidermal growth factor (EGFR) on cancer cells via a BsAb.
  Arms: Cohort 2 Arm A
Drug: EDV-GC — EDV-GC is a product based on the EnGeneIC EDV™ technology. EDVs are bacterially derived nanocells 400 nm in diameter that can be packaged with a range of different drugs. EDV-GC packages the immunomodulatory adjuvant aplha-galactosyl ceramide (GC) into the EDV and is designed to recruit anti-tumor immune cells.
  Arms: Cohort 2 Arm A
Drug: Gemcitabine — Gemcitabine in combination with nab-paclitaxel is routinely used as second-line therapy in metastatic PDAC patients who have either progressed on or are intolerant to 5-FU based combination in the first line setting. In this trial the safety and efficacy of E-EDV-D682/GC will be tested in combination with a reference therapy - gemcitabine and nab-paclitaxel.
Drug: Nab paclitaxel. — Nab-paclitaxel in combination with gemcitabine is routinely used as second-line therapy in metastatic PDAC patients who have either progressed on or are intolerant to 5-FU based combination in the first line setting. In this trial the safety and efficacy of E-EDV-D682/GC will be tested in combination with a reference therapy - gemcitabine and nab-paclitaxel.

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability and overall survival (OS) of E-EDV-D682/GC in combination with gemcitabine and nab-paclitaxel versus gemcitabine and nab-paclitaxel alone in participants with metastatic pancreatic ductal adenocarcinoma (PDAC) who have progressed on therapy.

DETAILED DESCRIPTION:
This study is testing an experimental treatment for participants with metastatic PDAC who have progressed following first line therapy involving 5-fluorouracil-containing combination that included irinotecan and oxaliplatin.

The experimental treatment consists of a chemotherapy drug, PNU-159682 packaged inside an EDV™ nanocell targeted to the epidermal growth factor receptor (EGFR) to form the investigational product E-EDV-D682. The EnGeneIC Dream Vector (EDV) nanocell is used to transport the chemotherapy directly to the tumor via the blood stream where it attaches to the surface of EGFR expressing cancer cells causing the cancer cells to die.

The E-EDV-D682 are given at the same time as one other investigational product designed to boost the body's own immune system to fight the cancer. This investigational product consists of non-targeted EDVs carrying alpha-galactosylceramide (GC) called EDV-GC. The combination of these 2 drugs is known as E-EDV-D682/GC.

The trial is a randomized blinded Phase I/IIa study that aims to test the safety and efficacy of E-EDV-D682/GC in combination with gemcitabine and nab-paclitaxel. The trial consists of 2 cohorts:

* Cohort 1 is an initial safety run-in phase that includes at least six participants who will receive E-EDV-D682/GC in combination with gemcitabine and nab-paclitaxel to assess safety. If one or less of the participants experience a dose limiting toxicity (DLT), the randomization portion of the study will be activated. If two or more DLTs occur, then the dose level will be reduced for the following participants. Cohort 1 enrollment will be complete once the first six evaluable participants have completed the DLT evaluation period, the study will then proceed to the randomized, blinded expansion phase.
* Cohort 2 is the randomized phase II expansion phase of the trial:

Participants will be randomized 2:1 to ARM A or ARM B, respectively:

1. ARM A. E-EDV-D682/GC with gemcitabine and nab-paclitaxel (N = 92)
2. ARM B. Gemcitabine and nab-paclitaxel with placebo (N = 46)

The first treatment cycle for all participants will involve bi-weekly visits for 3 weeks with a treatment free week in week 4, followed by weekly visits for a further 3 weeks. Doses of E-EDV-D682/GC in 3mL of 0.9% sodium chloride are administered intravenously over 10 seconds. In week 8, tumor burden will be radiologically re-evaluated in accordance with immune Response Evaluation Criteria in Solid Tumors (iRECIST) guidelines to determine treatment response.

Subsequent cycles will consist of weekly visits for 7 weeks. Following each 7-week treatment period is a treatment free week in which tumor burden is radiologically re-assessed (Week 8). Treatment may continue until the patient or investigator deems it suitable to stop treatment, for example if serious side effects occur or if the participants disease continues to grow.

It is estimated that the study duration for participants in the active treatment phase will be approximately 6 months consisting of two weeks for screening, 16 weeks of treatment (2 cycles, depending on the disease state and tolerability to the IMP and a 30-35-day safety follow-up visit).

ELIGIBILITY:
Inclusion Criteria:

* Histological or pathological confirmation of metastatic pancreas adenocarcinoma. Cytological or histological evidence of metastatic disease is required.
* Male or Female greater than or equal to 18 years of age.
* Eastern Cooperative Oncology Group (ECOG) performance score of 0-1.
* Life expectancy ≥ 3 months in the opinion of the Investigator.
* Measurable disease as per iRECIST criteria.
* Subjects must have tumors that express EGFR.
* Documented disease progression with first line FOLFIRINOX or NALIRIFOX therapy, during or within 3 months (+/- 15 days) after end of therapy.
* No more than one line of prior systemic therapy for metastatic PDAC allowed.
* Albumin level > 3.0 g/dl
* Adequate hematological function.
* Adequate renal function.
* Adequate hepatic function.
* Adequate cardiac function with LVEF ≥ 50% at baseline.
* Reproductive criteria as follows:
* Female subjects who are of non-reproductive potential
* Female subjects of childbearing potential must have a negative serum pregnancy test within 14 days of the first dose.
* Female subjects must be willing to use highly effective methods of birth control during the period of therapy and for 6 months following the last study drug administration.
* Male subjects must be willing to use highly effective methods of birth control during the period of therapy and for 6 months following the last study drug administration.
* All study subjects must be willing to ensure that corresponding sexual partners practice these same methods of highly effective birth control for the same duration.
* The subject (or subject's legally authorized representative) has provided voluntary signed informed consent.
* According to the investigator's assessment, subject will be able to comply with the study protocol.

Exclusion Criteria:

* Subjects currently receiving any other investigational agent.
* Unresolved (≥ Grade 1) non-hematological adverse events from prior anti-cancer therapy that is not controlled on maximal supportive therapy.
* Significant pericardial effusions, pleural effusions, or ascites that requires intervention. Subjects who require drainage within the last four weeks are ineligible.
* History of leptomeningeal or brain/CNS metastases.
* Ongoing treatment for other malignancies (hormone therapy acceptable).
* Patient may not have a history of malignancy other than PDAC within two years prior to screening except in circumstances where the risk of recurrence, metastasis or death in 5-years is <10%.
* Concurrent unstable diabetes mellitus or other contraindications for the use of corticosteroids that requires active titration of insulin.
* Subject has experienced a history of uncontrolled coronary artery disease, with or without angina pectoris or myocardial infarction, symptomatic congestive heart failure (New York Heart Association > Class II)
* Uncontrolled hypertension (systolic > 180 mmHg or diastolic > 100 mmHg) within two weeks.
* Uncontrolled cardiac arrhythmias requiring anti-arrhythmic therapy within the last four weeks.
* Baseline QTcF ≥ 450 ms (males) or ≥ 470 ms (females).
* Uncontrolled HIV infection. Patients without a prior diagnosis of HIV infection will undergo HIV testing unless not permitted to do so under local regulations. Patients with known HIV who have controlled infection (viral load undetectable and a CD4 count >350 either spontaneously or on a stable antiviral regimen) are permitted.
* Uncontrolled Hepatitis B virus (HBV) infection (chronic or acute).
* Uncontrolled Hepatitis C virus (HCV) infection.
* Uncontrolled arterial or venous thrombosis.
* Active or uncontrolled severe infection.
* Uncontrolled hypercalcemia (>2.6mmol/L or >10.3mg/dL) or symptomatic hypercalcemia requiring continued treatment for hypercalcemia.
* Received the following procedures within 21 days to receiving their first dose (or has not recovered from the toxic effects of such therapy) including:
* other investigational therapy
* radiotherapy
* any major surgery.
* Prior other therapies or procedures prior to receiving their first dose:
* QTc interval prolonging medicines should be reviewed and where possible their use should be minimized and alternate medicines that are not QTc interval prolonging, considered as substitutes.
* Known allergy/hypersensitivity to investigational components or excipients (trehalose, monoclonal antibody infusions, interferon therapy, or ciprofloxacin HCl (or other quinolones).
* Female who is pregnant or breastfeeding.
* Subject who cannot comply with protocol scheduled study visits or procedures, to the best of the subject and Investigator's knowledge.
* Any kind of disorder that, in the opinion of the Investigator, may compromise the ability of the subject to give written informed consent and/or to comply with all required study procedures.
* History or evidence of any other clinically significant disorder, condition, or disease (except for those outlined above) that, in the opinion of the Investigator would pose a risk to subject safety or interfere with the study evaluation, procedures or completion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2026-01-12 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment-Related Adverse Events as Assessed by CTCAE v5.0 | All adverse events will be monitored throughout the trial from the date of enrollment until 30 days after the last dose of study drug, on average 9 months.
  All participants will be monitored for adverse events (AEs) and serious adverse events (SAEs) according to the CTCAE (Common Terminology Criteria for Adverse Events), Version 5 criteria.
  Incidence and severity of AEs will be reported for individual participants and treatment arms. The safety of Gemcitabine Nab-paclitaxel + E-EDV-D682/GC (Arm A) will be compared to Gemcitabine Nab-paclitaxel + placebo (Arm B).
Duration of time from the start of treatment that participants are still alive. | Overall survival will be monitored from the date of first dose to the end of the treatment period (on average 9 months), then at 3 month intervals following discontinuation of study treatment for a minimum period of 12 months.
  A primary objective of the randomized, blinded Phase IIa stage of the study is to examine the overall survival rate for each treatment arm. i.e. Gemcitabine Nab-paclitaxel + E-EDV-D682/GC (Arm A), compared to Gemcitabine Nab-paclitaxel + placebo (Arm B). Overall survival is defined as time from the date of first administration of drug to the date of death, regardless of cause. Kaplan Meier curves will be utilized to determine percentage and median survival.
  The primary hypotheses that the IMP treatment improves overall survival versus standard-of-care chemotherapy will be assessed using statistical models defined in the study protocol.

SECONDARY OUTCOMES:
The number of days from the date of first administration of EDVs to the date of radiological evidence of disease progression | Imaging will be performed at baseline (screening) and at the completion of every cycle of treatment (8 weeks) until disease progression is confirmed by iRECIST or death, whichever comes first, up to 24 months.
  Progression free survival (PFS) will be calculated from all participants as the number of days from the date of first administration of EDVs to the date of radiological evidence of disease progression (date of MRI scan) or death, regardless of cause. A comparison of the PFS will be made between the two treatment Arms.
Percentage of participants with immune complete response (iCR) or immune partial response (iPR) | Imaging will be performed at baseline (screening) and at the completion of every cycle of treatment (8 weeks) until the participant is withdrawn from treatment (up to 24 months).
  The Objective Response Rate (ORR) will be measured as the percentage of participants with immune complete response (iCR) or immune partial response (iPR). A comparison of the ORR will be made between the two treatment Arms.
Time from initial response to disease progression | Imaging will be performed at baseline (screening) and at the completion of every cycle of treatment (8 weeks) until the participant has confirmed disease progression per iRECIST or death, whichever comes first, up to 24 months.
  The Duration of Response (DOR) will be measured as the time from the initial complete or partial response until disease progression or death, whichever comes first. A comparison of the DOR will be made between the two treatment Arms.
The proportion of participants with a disease response at 4 months after treatment initiation | Imaging will be performed at baseline (screening) and at the completion of cycle 2 of treatment (16 weeks).
  The Disease Control Rate (DCR) will be measured as the proportion of participants with immune complete response (iCR), immune partial response (iPR) and immune stable disease (iSD) at 4 months after treatment initiation. A comparison of the DCR will be made between the two treatment Arms.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Linda Y.Wu, MD, Principal Investigator — Columbia University Medical Center/ Herbert Irving Pavilion; Dr Jennifer MacDiarmid, Ph.D, Study Director — Engeneic Pty Limited; Dr Himanshu Brahmbhatt, Ph.D, Study Director — Engeneic Pty Limited
Locations (3):
- United States (3):
  - Atlantic Health, Summit, New Jersey
  - Columbia University Irving Medical Center, New York, New York
  - Taylor Cancer Center, Maumee, Ohio

IPD SHARING:
Plan to Share IPD: No